CLINICAL TRIAL: NCT03726983
Title: Randomized Controlled Trail of e-Health Management for Women With Prior Gestational Diabetes Mellitus
Brief Title: The Effect of E-Health Management on Gestational Diabetes Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Mei-Chen Su, Director, Clinical Research, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 105-4129C
Record Dates: First submitted 2018-10-29; First posted 2018-11-01 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy
Keywords: gestational diabetes mellitus; pregnant women; e-health management; metabolic syndrome
MeSH Terms: conditions — Diabetes, Gestational; Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: This study was longitudinal approach and repeated testing using an experimental design to evaluate the follow-up outcomes of the e-heath management platform intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eHMP experimental group (Experimental): The experimental group received health management support and counseling,including:
  1. GDM health care knowledge
  2. self-awareness of health
  3. self-monitoring of health status (i.e., recording weight and measurement data of metabolic syndrome risk factors and monitoring changes in data trends)
  4. participation in discussions or browsing forums
  5. healthy lifestyle guidance and counseling
  6. reminder systems
  7. a token system of earning points in exchange for prizes.
  Interventions: Other: Experimental group
- Control group (No Intervention): only received usual care

INTERVENTIONS:
Other: Experimental group — Pregnant women who agree to take part will be assigned to a group: experimental group and control group. The experimental group will received health management support and counseling that were conducted by the researchers through the e-health management platform.
  Other Names: e-Health Management Platform
  Arms: eHMP experimental group

SUMMARY:
The purpose of this study was to develop an e-heath management platform(eHMP) for women with high risk of gestational diabetes mellitus (GDM) and to evaluate the longitudinal effects between groups of eHMP intervention.

DETAILED DESCRIPTION:
Background: Women with previous gestational diabetes mellitus are at increased risk for developing type2 diabetes mellitus or metabolic syndrome in their later life. Infants of mothers with GDM are more susceptible to stillbirth and more serious health concerns. With limited time for visits and the predicament of education, applying web-based intervention has become a convenient tool for health management.

Objectives: The approved project aimed to develop an e-heath management platform(eHMP) for women with high risk of gestational diabetes mellitus (GDM) and to evaluate the longitudinal effects between groups of eHMP intervention. The eHMP integrate GDM health care knowledge, self-awareness of health, self-monitoring of health status (i.e., recording weight and measurement data of metabolic syndrome risk factors and monitoring changes in data trends); participation in discussions or browsing forums; healthy lifestyle guidance and counseling; reminder systems, a token system of earning points in exchange for prizes.

Methods: Pregnant women aged 18-45 years with high risk of metabolic syndrome who have a singleton pregnancy, are eligible to participate in this study. Women who agree to participate in the study will be given a participant information sheet and consent form. Participants will be recruited from the Pregnancy diabetes Clinic, at Chang Gung memorial hospital and introduced to the eHMP using the mobile phone in the clinic. Participants will also be given the URL to access to the program and they can learn the modules at home by using their home PCs, mobile phones, or tablets. They were followed up for three times: 28 weeks' gestation, 36-40 weeks' gestation and 6-12 weeks postpartum. SPSS version 20.0 software was used to compile and analyze the research data, including questionnaires and blood test for metabolic index.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women (pre-pregnancy body mass index ≧ 24) must meet at least one of the following conditions and agree to be interviewed:

* Age over 34 years old;
* Ever had giant infant delivery (weight ≧ 4.5 kg);
* Previous diagnosed with gestational diabetes ;
* Family history of diabetes.

Exclusion Criteria:

* Pre-existing diabetes (types 1 and 2);
* Unable to write and understand Chinese;
* Subject has cognitive impairment;
* Subject has intellectual disability or mental illness;
* Dependent on medical care (eg, anti-depressants, or any psychiatric medication)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2017-01-05 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Change of Triglyceride Level | Change from Baseline at 6-12 weeks after delivery
  Blood sampling was performed in the fasting state. Normal triglyceride was <150 mg/dl; ≥150mg/dl was abnormal
Change of Fasting Blood Glucose (FBG) Level | Change from Baseline at 6-12 weeks after delivery
  Blood sampling was performed in the fasting state. Normal FBG was < 100 mg/dl; ≥100mg/dl was abnormal
Change of high-density lipoprotein cholesterol (HDL) level | Change from Baseline at 6-12 weeks after delivery
  Blood sampling was performed in the fasting state. Normal HDL was ≥50 mg/dl; <50mg/dl was abnormal
Change of Cholesterol level | Change from Baseline at 6-12 weeks after delivery
  Blood sampling was performed in the fasting state. Normal Cholesterol was < 200 mg/dl; ≥200mg/dl was abnormal
Change of systolic blood pressure | Change from Baseline at 6-12 weeks after delivery
  Normal systolic blood pressure was <130mmHg; ≥130mmHg was abnormal. Blood pressure was measured at the right arm twice after a 10-min rest in the supine position by using a calibrated sphygmomanometer and averaged.
Change of diastolic blood pressure | Change from Baseline at 6-12 weeks after delivery
  Normal diastolic blood pressure was <85mmHg; ≥85mmHg was abnormal. Blood pressure was measured at the right arm twice after a 10-min rest in the supine position by using a calibrated sphygmomanometer and averaged.
Change of body weight | Change from Baseline at 6-12 weeks after delivery
  Women's weight following as assessed using calibrated digital scales
Newborn baby weight | at birth
  Newborn baby weight in normal range (>2500g - <4500g) - dichotomous outcome Yes/No assessed using calibrated digital scales.

SECONDARY OUTCOMES:
Change of Pregnancy Physical Activity Assessment | Change from Baseline at 6-12 weeks after delivery
  There are 12 items in this questionnaire, including two dimensions: exercise and inactivity. Exercise dimension contained four items to assess the type of physical activity, intensity, duration, frequency during pregnancy. At least 3 days per week, and each time at least 20-30 minutes, counted as regular exercise (dichotomous outcome Yes/No assessed). Inactivity dimension contained 8 items, dichotomous outcome Yes/No assessed (score 0-8), higher values represent an inactivity lifestyle.
Change of Dietary Behavioral Characteristics Scale | Change from Baseline at 6-12 weeks after delivery
  The instrument is 17-item Likert-type self-report instrument, used a 5-point response format to obtain data regarding the frequency of reported behaviors (never, rarely, sometimes, usually, always). It including two dimensions and each scale range as: balanced diet (5 items, scale range 5-25) and diet control behavior (12 items, scale range 12-60). Higher values represent a better maternal dietary patterns during pregnancy.
Change of Health Promotion Scale | Change from Baseline at 6-12 weeks after delivery
  The instrument is 40-item Likert-type self-report instrument, used a 5-point response format to obtain data regarding the frequency of reported behaviors (never, rarely, sometimes, usually, always). It including six dimensions and each scale range as: social-support (6 items, scale range 6-30), life-appreciation (8 items, scale range 8-40), health-responsibility (8 items, scale range 8-40), stress-management (9 items, scale range 9-45), nutritional behaviors (5 items, scale range 5-25) and exercise behaviors (4 items, scale range 4-20). The total score was 40 to 200, higher values represent a better health promotion lifestyle.

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Chen Su, Dr., Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorail Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No